CLINICAL TRIAL: NCT01623908
Title: An Open,Multicentre,Prospective Study of Adjuvant Zoledronate Treatment in Osteoporosis Women With Breast Cancer
Brief Title: Bone Loss Treatment From Adjuvant Zoledronate Efficacy
Acronym: BLAZE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Lin, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110618GD
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasms; Bone Loss
Keywords: Breast neoplasms; Zoledronate; Bone loss
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases, Metabolic | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronate (Experimental)
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Zoledronate — 4mg, IV (in the vein) every 6 months. Number of Cycles: up to the researcher or until unacceptable toxicity develops.
  Other Names: Zometa

SUMMARY:
The main purpose of this study is to observe and assess the impact of adjuvant zoledronate on bone density in breast cancer patients.

The second purposes:

* The efficacy of adjuvant zoledronate
* The safety of adjuvant zoledronate
* The bone loss of breast cancer patients in Guangdong
* The correlation between bone loss of breast cancer patients and treatment of disease in Guangdong

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed malignant disease and the leading cause of cancer-related mortality among women.

Zoledronate is a bone-targeted bisphosphonate, which is used to treat osteoporosis and to reduce the risk of skeletal morbidity in patients with bone metastases. Zoledronate can also reduce the persistence of disseminated tumour cells in the bone marrow of women with early-stage breast cancer. Nowadays, consensus is emerging that certain subsets of patients with early-stage breast cancer may benefit from bisphosphonate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female, age > 18.
* Postoperative breast cancer patients who have finished adjuvant chemotherapy or unwilling to receive chemotherapy.
* T score < -2.0, or -2.0 < T score <-1.0 with any 2 of the following risk factors: T score < -1.5, age > 65, BMI < 20kg/m^2, family history of hip fractures, age > 50 with brittle fracture history, oral steroid therapy > 6 months, receiving aromatase therapy.
* ECOG(Eastern Cooperative Oncology Group) physical state score:0-2.
* Breast cancer stage I-III confirmed by histological or cytological examination.
* Patients received radical surgery with estimated survival time > 12 months.
* Laboratory tests should be performed 1 week before enrollment and the results should meet the following criteria: neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 100×10^9/L, hemoglobin ≥ 80g/L, serum bilirubin ≤ 1.0×ULN, AST and ALT ≤ 1.5×ULN, Serum creatinine ≤ 1.0×ULN.
* Patients who never received intravenous bisphosphonate within 12 months before enrollment and did not receive oral bisphosphonate within 3 weeks before enrollment.
* Informed consents should be signed by the participants or their guardians. All the participants should be aware of the purpose and procedure of this study and willing to participate in this study.
* Contraception required for those reproductive-aged women.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients who have not signed informed consent.
* Patients received medical treatment which can affect bone metabolism (such as calcitonin, mithramycin or gallium nitrate) within 2 weeks before enrollment.
* Bone metabolic diseases such as Paget's disease, epiphyseal dysplasia and primary or secondary hyperthyroidism diagnosed within 12 months before enrollment.
* Liver function impairment which is defined as 2.5-fold or more increase in ALT or AST levels compared with the upper limit of reference range.
* Refuse appropriate contraception (appropriate contraceptive options include female sterilisation, intrauterine device, oral contraceptives and barrier contraception).
* Active dental diseases including dental infection, mandibular pain and maxillary or mandibular trauma. Patients with mandibular osteonecrosis diagnosed currently or previously, exposed bone or slow healing after oral surgery. Patients who will receive dental or maxillofacial surgery (such as dental extraction and dental implant) in the first 6 weeks after enrollment.
* Patients with dysgnosia or communication disorder who can't well understand our study, cooperate with our staff or operate glucose monitor correctly.
* Combined with major organ dysfunction or other severe diseases such as severe coronary disease, cardiovascular disease, myocardial infarction occurred within 12 months before enrollment, severe neurological or psychiatric diseases, severe infection or active disseminated intravascular coagulation.
* Alcoholics or drug addicts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Bone Mineral Density | 48 weeks

SECONDARY OUTCOMES:
Bone metastasis rate | From date of randomization until the date of bone metastasis, assessed up to 48 weeks.
Disease-Free Survival | From date of randomization until the date of bone metastasis or date of death from any cause, whichever came first, assessed up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shenming Wang, MD, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University; Ying Lin, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (10):
- China (10):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - GuangDong Hospital Of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Shenzhen Second Municipal People's Hospital, Shenzhen, Guangdong